CLINICAL TRIAL: NCT07004998
Title: Comparison of Left Paratracheal Versus Cricoid Pressure on Glottic Visualization During Videolaryngoscopy: A Randomized Crossover Study
Brief Title: PARAtracheal vs CRIcoid Pressure on GLIttic DEformation (PARAGLIDE)
Acronym: PARAGLIDE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Benjamin Javillier, MD, Principal Investigator, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PARAGLIDE
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Airway Management
MeSH Terms: interventions — N 30

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Pressure (Baseline) (No Intervention): Videolaryngoscopy performed without any external laryngeal pressure. This serves as the baseline condition for each patient.
- Cricoid Pressure (30 N) (Active Comparator): Videolaryngoscopy performed while applying standardized cricoid pressure (30 N) by a trained operator. A video image is captured during this maneuver.
  Interventions: Procedure: Cricoid Pressure (30 N)
- Left Paratracheal Pressure (30 N) (Experimental): Videolaryngoscopy performed while applying standardized left paratracheal pressure (30 N) by the same operator. A video image is captured during this maneuver.
  Interventions: Procedure: Left Paratracheal Pressure (30 N)

INTERVENTIONS:
Procedure: Cricoid Pressure (30 N) — Manual application of posterior pressure on the cricoid cartilage at a standardized force of 30 newtons. The pressure is applied by a trained operator using one or two fingers, with the goal of compressing the esophagus against the cervical spine. The maneuver is performed after induction of general anesthesia and immediately before videolaryngoscopy. A still image of the glottic view is captured during pressure application.
  Other Names: Sellick Maneuver; Cricoid Force; CP; Cricoid Compression; Cricoid Pressure
  Arms: Cricoid Pressure (30 N)
Procedure: Left Paratracheal Pressure (30 N) — Manual application of pressure to the left paratracheal region, lateral to the trachea and inferior to the thyroid cartilage, at a standardized force of 30 newtons. The pressure is applied by a trained operator using the thumb or fingers. The maneuver is performed after induction of general anesthesia and immediately before videolaryngoscopy. A still image of the glottic view is captured during pressure application.
  Other Names: LPP; Left Paratracheal Pressure
  Arms: Left Paratracheal Pressure (30 N)

SUMMARY:
This randomized crossover study evaluates the effects of left paratracheal pressure, cricoid pressure, and no pressure on glottic visualization during videolaryngoscopy in adult surgical patients. The primary endpoint is the Percentage of Glottic Opening (POGO) score assessed by blinded video review. Secondary endpoints include anatomical measures (glottic surface area, vertical and horizontal displacement of the glottic plane) and clinical outcomes (first-pass success, first-pass success without desaturation <90%, intubation time, Intubation Difficulty Scale, hypoxemia, hemodynamic events, airway trauma, and postoperative sore throat or dysphonia). All outcomes are collected from routine anesthetic practice and video analysis, with no additional procedures.

DETAILED DESCRIPTION:
This randomized crossover trial will compare three laryngoscopy conditions (no pressure, cricoid pressure, left paratracheal pressure) in adult surgical patients requiring general anesthesia with tracheal intubation. Each patient undergoes all three conditions in random order, with the intubation performed using the maneuver chosen by the operator. Anatomical outcomes (POGO, glottic surface area, vertical and horizontal displacement of the glottic plane) will be assessed from video recordings by blinded evaluators. Clinical outcomes (first-pass success, composite success without desaturation <90%, intubation time, IDS, hypoxemia, hemodynamic changes, airway trauma, sore throat, dysphonia) will be collected from routine anesthetic records and PACU assessments.

Statistical Analysis Plan:

POGO: mixed-effects repeated measures model with patient as random effect, maneuver as fixed effect, adjusted for operator, BMI, and Mallampati.

Anatomical outcomes: analyzed similarly with mixed models and planned contrasts (LPP vs CP).

Clinical outcomes: analyzed as-treated, using logistic or linear regression with adjustments for baseline factors and operator as random effect.

Mediation analysis will evaluate whether improvements in POGO explain clinical benefits (first-pass success, intubation time).

Significance level set at α=0.05 (two-sided), with exploratory outcomes interpreted without multiplicity correction.

Missing data (e.g., unusable videos, missing sore throat scores) will be reported; complete-case analysis will be primary, sensitivity analysis considered if >5% missing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled for elective surgery under general anesthesia requiring endotracheal intubation
* ASA physical status I or II
* Normal airway anatomy as assessed by the anesthesiologist (Mallampati I-II, no known or anticipated difficult airway)
* Written informed consent obtained prior to inclusion

Exclusion Criteria:

* History of difficult intubation or anticipated difficult airway
* Known upper airway anatomical abnormalities (e.g., tumors, tracheal deviation, cervical spine instability)
* BMI > 35 kg/m²
* Gastroesophageal reflux disease or increased aspiration risk
* Pregnancy
* Emergency surgery
* Allergy or contraindication to any anesthetic drugs used
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Glottic Opening (POGO) score | During laryngoscopy, before tracheal intubation
  POGO will be scored from video recordings of each condition (no pressure, cricoid, paratracheal) by blinded assessors (0-100%).

SECONDARY OUTCOMES:
Glottic surface area | During laryngoscopy, before intubation
  Glottic surface area will be quantified from videolaryngoscopic images under each condition (no pressure, cricoid, paratracheal) using standardized image analysis by blinded reviewers.
Vertical Displacement of the Glottic Plane | During laryngoscopy, before intubation
  The vertical shift of the glottic plane relative to baseline will be measured on recorded videolaryngoscopic images under each condition, assessed by blinded reviewers.
Horizontal displacement of the glottic plane | During laryngoscopy, before intubation
  The horizontal (lateral) shift of the glottic plane relative to baseline will be measured on recorded videolaryngoscopic images under each condition, assessed by blinded reviewers.
First-pass intubation success | From laryngoscope insertion to first confirmed capnography
  Successful tracheal intubation at the first attempt with the maneuver chosen by the operator.
Time to intubation | From laryngoscope insertion to first confirmed capnography
  Duration in seconds until successful tracheal intubation.
Intubation Difficulty Scale (IDS) | During intubation
  Composite score including attempts, operators, optimization maneuvers, and force required.
First-attempt success without desaturation < 90% | From laryngoscope blade past the incisors until confirmed tracheal intubation (end-tidal CO₂ ≥ 5 mmHg for 3 breaths), typically up to 2 minutes.
  Binary composite. Success = both (1) first-attempt intubation (tube placed without complete blade removal; optimizations allowed without blade withdrawal) and (2) no SpO₂ < 90% for ≥ 5 s within the time frame.
Hypoxemia | From induction until confirmed intubation
  Oxygen saturation <92% recorded by pulse oximetry.
Hemodynamic events | From induction until confirmed intubation
  Systolic blood pressure drop >20% from baseline or heart rate <50/min.
Airway trauma | Immediately after intubation
  Blood on blade/stylet or visible lip/mucosal injury.
Postoperative sore throat | 30-60 minutes in PACU
  Patient-reported throat pain on numeric scale (0-10).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint-Luc, Bouge, Namur, Belgium

IPD SHARING:
Plan to Share IPD: Yes
What: de-identified outcome data (clinical and imaging) and analysis code; selected de-identified video frames. When: after publication. How: upon reasonable request to the sponsor/PI with data-use agreement.